1.1

# Patient-Clinic-Community Integration to Prevent Obesity Among Rural Preschool Children (ENCIRCLE)


#### **Abbreviations:**

**AAP - American Academy of Pediatrics** 

BMI - Body Mass Index

EHR - Electronic Health Record

FNPA - Family Nutrition and Physical Activity

IRB - Institutional Review Board

**ISO – Information Security Office** 

IT - Information Technology

PACO – Patient Advisory Council on Obesity

**PCP – Primary Care Provider** 

**PRO – Patient-Reported Outcome** 

SNAP-Ed - United States Department of Agriculture's Supplemental Food and Nutrition Assistance Program-Education

WCV - Well Child Visit

Encircle Protocol Version 1.21 Version Date: 11/29/2022

IRB #: 2020-0207

#### INTRODUCTION

A proliferation of family-based interventions have been developed to prevent (and treat) childhood obesity, yet only one systematic review has examined the effectiveness of preventive interventions by delivery setting. 11 This review of 139 prevention intervention studies showed that 83% were primarily school-based and provided support for a multi-level environment approach that included school, home, and community components. 11 However, evidence through 2013 was insufficient for *non-school* based interventions, thus offering no clear direction for obesity prevention for preschool-aged children. 11 Likewise, a qualitative content analysis 43 of 119 prevention studies from 2008 to 2015 reported that only 1 in 5 studies used a multi-level setting approach, and none compared the effectiveness of varied levels, further underscoring the gap regarding the need to understand the comparative effectiveness of preventive care models for preschool-aged children. This project responds to this gap by comparing the relative effectiveness of clinic, patient-clinic, and patient-clinic-community interventions to prevent obesity among preschool-aged children in rural, low-income families at high risk for obesity.

#### **BACKGROUND AND RATIONALE**

Magnitude and Persistent Health Burden of Child Obesity: In 2018, more than 2 million US children began kindergarten with obesity. 12 The US prevalence of obesity among preschoolaged children increased from 10.1% in 2007-2008 to 13.9% in 2015-2016.30 Low family income and community-level socio-economic deprivation in childhood increase risk for obesity and overweight through adolescence.<sup>27,31</sup> Rural residency is also associated with higher body mass index (BMI) in childhood and increased odds for childhood obesity. 12-15 Practitioners and policy makers are cognizant of this disparity, yet rural children remain underrepresented in the literature. The preschool years are a critical period for preventive interventions as rapid gains in BMI during this period lead to early-life obesity and a substantial health burden during childhood, including poor cardiovascular and metabolic health characterized by high blood pressure, dyslipidemia, and insulin resistance, 32-35 and other adverse physical health effects such as asthma, obstructive sleep apnea, early maturation, polycystic ovarian syndrome, and nonalcoholic hepatic steatosis. 36,37 Further, children with obesity report adverse social and emotional health including lower self-esteem and health-related quality of life compared to children with normal weight status.<sup>38</sup> These effects during childhood are certainly problematic, but the primary public health burden is the persistence of obesity and duration of adverse effects over time. Longitudinal studies indicate that 60 to 90 percent of preschool-aged children with obesity had persistent obesity into adolescence<sup>2,3</sup> and adulthood.<sup>39</sup> Obesity that persists into adulthood has detrimental effects on health, with a significant impact on population health: based on the prevalence of obesity among children aged 2-19 years in 2016, and assuming no gains in secular trends, 57% of the US population is expected to be obese by age 35 years and will face serious co-morbidities.40

Rationale for targeting preschool children: Preschool children are the focal population for this project to respond to a scientific gap in understanding the comparative effectiveness of preventive intervention strategies for preschool-age children. Obesity prevention may have the greatest preventive benefit if begun early in life, before age 2 years, and there is an opportunity to meet patients where they are in clinical well child visits (WCVs) and to extend care in


Encircle Protocol Version 1.21 Version Date: 11/29/2022 IRB #: 2020-0207 community settings.<sup>41</sup> Risk factors for early childhood obesity may include maternal prepregnancy BMI, excessive gestational weight gain, curtailed infant sleep, and inappropriate bottle use among other factors<sup>42</sup> whereas the Family Nutrition and Physical Activity (FNPA) patient-reported outcome (PRO) screening tool is appropriate for assessing risk factors observed in preschool children (e.g., snacking, organized play).

**PCP Roles and Responsibilities:** The primary care provider (PCP) is the central actor in the clinic setting and responsible for adopting clinical guidelines<sup>9,10</sup> for obesity prevention that include BMI screening, behavioral risk assessment (nutrition, physical activity, sedentary activity, sleep), and delivering individually-tailored, family-centered preventive counseling. PCPs face decisional dilemmas that hinder adoption of these clinical guidelines,<sup>44</sup> with three major gaps identified: 1) what tool to use to assess behavioral risk for obesity;<sup>9,44</sup> 2) how to meet parent expectations for individually-tailored, family-centered preventive counseling that meets children's developmental needs;<sup>9,10,20</sup> and 3) the unknown efficacy of guideline implementation on obesity prevention.<sup>10,11</sup> The comparators address these gaps, thereby assisting PCPs in determining how best to counsel parents of preschool-aged children at risk of obesity.

FNPA Behaviors Targeted: There is general consensus that effective obesity prevention should target: 1) poor diet (e.g., consumption of sugar-sweetened beverages and energy-dense foods); 2) low levels of physical activity; 3) short sleep duration; 4) sedentary behaviors (e.g., high media use); and 5) parenting practices. 45-49 Only 16% of 119 studies reviewed in a qualitative content analysis 43 of obesity prevention studies adhered to guidance recommending that all behaviors be addressed, with media use and sleep being under-addressed. The FNPA PRO measure and risk assessment addresses all 5 behaviors (Appendix A) and is a valid clinical tool to identify risk factors associated with obesity 50-52 among preschool-aged children and related chronic disease indicators (adiposity measures, severity of obesity, cardiovascular disease risk, and glucose intolerance). 53-55 The FNPA risk assessment offers time efficiencies to clinicians as parents self-assess risk to allow the PCP to focus discussion on relevant, family-centered issues.

**Food Insecurity**: A majority of childhood obesity prevention studies have targeted populations with low-income but no interventions included in recent systematic reviews<sup>11,43,56-58</sup> have addressed food insecurity, a well-recognized moderator of obesity. 59-62 In fact, a 2018 randomized controlled trial of parents of preschool-aged children who received all 5 behavioral targets in home and community settings failed to observe differences in BMI at 3 years followup except among families who were food insecure at baseline. 63 The American Academy of Pediatrics (AAP) issued guidance recommending food insecurity screening; this is a standard social determinant of health indicator in electronic health record (EHR) systems and fully implemented at Geisinger. <sup>64</sup> Professional guidance highlights the role PCPs play in referring families with food insecurity to community food access resources. Recent studies evaluating the feasibility and acceptability of PCPs in this role has emphasized the importance of providing PCPs with resources to facilitate referrals and ultimately empower parents to improve food security. 65-67 Geisinger PCPs have been asked to take action by referring pediatric patients and their parent(s) to Geisinger Wellness' collaborative effort with the Central Pennsylvania Food Bank in response to heighted food insecurity during the COVID-19 pandemic. Specifically, lost wages due to job layoffs and industry closures and limited availability of food due to shortages will strain households that were food insecure while other households will become newly food insecure. Changes in food security will be evaluated as a secondary outcome across all arms.

The specific aims for this project are follows:

- 1. To compare the effectiveness of WCV vs. PRO WCV vs. PRO WCV + Food Care on obesity prevention for preschool-aged children from rural, lower income households with BMI-forage and -sex > 50th percentile at baseline.
  - 1a. To examine the effectiveness of the interventions on the change in BMI z-score at 1-year follow-up, and on the percent of children overweight (> 85th percentile BMI-for-age and sex) and obese (> 95th percentile BMI-for-age and -sex) at 1-year.
  - 1b. To examine the effectiveness of the interventions on a secondary outcome related to parents' perceptions of being involved with the PCP in preventive counseling.
  - 1c. To examine the effectiveness of the interventions on secondary outcomes related to home and parent factors, including food resource management and household food security.
- 2. To examine multi-level mediators and moderators of effectiveness of each intervention.
  - 2a. To evaluate whether intervention effectiveness is mediated by parent and PCP attitudes, norms, perceived behavioral control and intention to prevent obesity.
  - 2b. To evaluate whether intervention effectiveness is mediated by child behaviors including nutrition, physical activity, screen time, and sleep.
  - 2c. To explore whether intervention effectiveness is moderated by community, clinic, and home factors. Community factors include socio-economic deprivation, rurality, and parents' perception of their neighborhood. Clinical organizational climate and household income and transportation will be evaluated.
- To identify factors influencing effective implementation at the parent, PCP, and clinic levels.
   To identify factors influencing parent completion and PCP utilization of the PRO measure.
  - 3b. To identify factors influencing use of family-centered preventive counseling.
  - 3c. To identify factors influencing parent utilization of community referrals.

#### **PROCEDURES**

#### Research Design

A cluster-randomized controlled trial will compare effectiveness of the two interventions (Arms 2 and 3) versus control (Arm 1) on the prevention of obesity among preschool-aged children (Aim 1). Geisinger PCPs who conduct WCVs (pediatricians, family or community medicine physicians, nurse practitioners) will represent the units of randomization (i.e., clusters). Families (the eligible child and their parent)—representing the individuals to which study findings will be generalizable—will receive one of the three interventions based on the comparator assignment of the PCP who conducts the child's WCV. Participating PCPs will be randomized into an intervention arm, which entails having changes made to their EHR interface and having these changes impact all preschool-aged children for whom they provide WCV (Arms 2 and 3). The EHR changes are novel to the eligible PCPs. Families will be consented to participate in the study follow-up, but not to the interventions, which require implementation on a system level. Cluster, rather than individual-level, randomization is warranted because of the automated EHR-based intervention, because PCPs cannot be expected to change their standard


Encircle Protocol Version 1.21 Version Date: 11/29/2022 IRB #: 2020-0207 clinical practices on a patient-by-patient basis, and because their obesity-prevention practices will likely be influenced by their exposure to FNPA (i.e., "contamination" concerns). The cluster design isn't without disadvantages. This design has the potential for imbalance of the number of subjects across PCP resulting in possible imbalance at the intervention level. Also, analyses are complicated with a small number of clusters (<20). To overcome these disadvantages, we have compensated for potential imbalance in the sample size calculations. Lastly, our chosen method of analysis appropriately handles imbalance and combined with a large number of clusters, a total of 60, we do not anticipate concerns in the implementation and analysis.

A stratified design will be used to reduce the imbalance of covariate distributions between intervention arms. Prior to randomization, PCPs will be stratified based on the type of clinic in which they practice (Pediatrics versus Community Medicine) and case load (number of annual WCV conducted among the target population; low volume (< 52 WCV/year) or high volume > 52 WCV/year), as heavy patient volume can disrupt workflow and may affect intervention delivery. 99,100 Since stratification can only address a limited number of potential confounders, initial analyses will examine other covariates known to influence clinical interventions and/or childhood obesity such as parent BMI, child baseline weight status, biological sex and race/ethnicity.

CORRECTION: Per discussion with the study team and PCORI in October 2022, it was observed that stratification details are an error. Per study documents, in August 2020 the study team observed that all but one pediatrician had a volume <52 WCVs in 2019, the past year, and Year-to-Date assessments; conversely, all Community Medicine providers had <52 WCVs. Therefore, 2 strata characterized: Pediatricians and Community Medicine. The Community Medicine providers were further stratified by those with <32 WCVs/year and those with >=32 WCVs/year to align with clinic eligibility criteria: "Eligible clinics will have  $\geq$ 1 PCPs with at least 32 qualifying well child visits annually for children aged 20 to 60 months,  $\geq$ 50th BMI-forage and -sex percentile."

Following randomization, PCPs' assignment to 1 of the 3 comparators will be revealed to PCPs. However, PCPs will be blind to whether individual patients are participating in the study follow-up. For Arm 3, post-WCV referrals to Food Care will be aided by a research assistant (not blind to PCP assignment) who will discuss the education program option with enrolled participants and document the referral in the child's EHR. Thus, at the point of the enrolled patient's baseline WCV, all PCPs will be blind to participant identity; only at follow-up visits will PCPs be aware of who is enrolled in Arm 3. Per practice guidelines and insurance schedules, WCVs are scheduled at >12-month intervals; however, children could return in the interim for acute care and a PCP may observe a child's prior exposure to a group through progress notes. Theoretically, the PCP providing acute care could "contaminate" the parent-child dyad by discussing healthy lifestyle behaviors, but pragmatically, the contamination risk is low due to high likelihood of maintaining care with the PCP who provided the WCV and low likelihood of a PCP discussing such behaviors during acute care visits (based on PCP and parent reports). Nonetheless, progress notes from child participants' EHR will be monitored over the study period to fully capture the dose of preventive counseling. To further reduce bias, study investigators, biostatisticians, and the project coordinator (responsible for collecting study questionnaires) will be blind to PCPs' intervention assignment. The project manager and data analyst will not be blind to intervention assignment, due to participant and data management responsibilities.

### **Study Population**

Human subjects include Geisinger pediatric patients, and their parents/caregivers, from Geisinger Pediatric and Community Medicine clinics. Human subjects also include Geisinger Pediatric and Community Medicine providers who meet study threshold for volume of annual well child visits.

Inclusion criteria for child participants include:

• Age (20-months to 59-months, 29-days old)

If the child is <24 month of age, then eligible if greater than or equal to 50th percentile for BMI-for-age and -sex at any visit (WCV, acute, etc.) since age >12 months or at enrollment.

If child is > 24 or <27 months of age, then eligible if greater than or equal to 50th percentile for BMI-for-age and -sex at any visit (WCV, acute, etc.) in the prior 12 month period or at enrollment.

If child is >27 months or <60 months of age, then eligible if greater than or equal to 50th percentile for BMI-for-age and -sex at any visit (WCV, acute, etc) in the prior 15 month period or at enrollment.

This study uses the World Health Organization (WHO) growth standards for inclusion criteria and the primary outcome, BMI z-score (https://www.who.int/childgrowth/standards/en/).

- Parent commitment to participate in 18-month study
- Plans to attend scheduled WCV and recommended follow-up WCV in 12 months
- No plans to move or change health systems in 2 years
- Parent age  $\geq$  18 years
- Parent is English-speaking
- Household is considered lower-income (i.e., eligible for or receiving Special Supplemental Nutrition Program for Women, Infants and Children [WIC], Supplemental Nutrition Assistance Program [SNAP], Temporary Assistance for Needy Families [TANF], Medicaid, or Children's Health Insurance Program [CHIP]), screens positive for food insecurity, National School Lunch or Breakfast participation, has picked up school lunch or breakfast at curbside during coronavirus, or has experienced job disruption due to coronavirus.

#### Child exclusion criteria include:

- Children who attend their regularly scheduled WCV via telemedicine
- Another child in family is participating
- Pre-existing medical exclusions (cancer, type 1 diabetes, major developmental delays such as autism)
- Parents with self-reported major depression will be excluded

Potentially eligible child patients will be initially screened and identified using an Electronic Health Record guery for patients meeting the study inclusion/exclusion criteria. Potentially eligible participants will also be screened in-person when they present at clinic for care; by

phone interview if the child has a scheduled well child visit but does not have an established history in the electronic health record (e.g., new patient); or online self-screening initiated by the parent/guardian (i.e., in response to seeing recruitment flyer, MyGeisinger message, social media ad, etc.).

#### **Participant Enrollment**

**Table 1**. Projected Enrollment

| Tuble 1. 1 Tojected Emonment | |
|---|---|
| 1. Estimated number of potentially eligible study participants (determined by Electronic Health Record): | 5,438 |
| 2. Total number of study participants expected to be screened: | 5,438 |
| 3. Total number of study participants expected to be eligible of those screened: | 3,643 |
| 4. Target sample size (use same number stated in milestones): | 2,025 |
| 5. If applicable, total number of providers that will enroll participants: | 100 |
| 6. Projected month first participant enrolled (month after project initiation): | Month 8 |
| 7. Projected month last participant enrolled (month after project initiation): | Month 35 |
| 8. Projected rate of enrollment (anticipated number enrolled per month of enrollment period): | 169 |
| 9. Estimated percentage of participant dropout: | 10% |

### **Study Procedures**

Geisinger Community Medicine and Pediatric Service Line leadership will attest to the inclusion of clinic sites to engage in the study. Eligible clinics will have ≥1 PCPs with at least 32 qualifying well child visits annually for children aged 20 to 60 months, ≥50<sup>th</sup> BMI-for-age and -sex percentile. Geisinger PCPs who qualify for participation in this research will be informed of the study asked to participate in a FNPA training (in-person and via Microsoft TEAMS) and complete study questionnaires referenced in **Appendix B** (clinic and PCP items). Baseline questionnaires will be self-administered and collected via hard copy (at training) or via RedCAP (following TEAMS training). For the purpose of implementation evaluation, PCPs will also be asked to complete follow-up questionnaires at 12 and 20 months; questionnaires will be administered via RedCAP. Attendance at a training session will be seen as implied consent to participate in the research.

Randomization will occur at the PCP level. PCPs in Arm 1 will be asked to provide usual well child visits. PCPs in Arms 2 and 3 will be asked to provide standard well child visits at Geisinger which include the FNPA screening tool. FNPA has been recognized as standard of care in some Pediatrics and Community Medicine clinics since 2013. FNPA implementation at Geisinger has occurred in phases to gradually scale-up and simultaneously allow for rigorous testing of efficacy and effectiveness. In this study, PCPs in Arm 1 will be considered "wait-list" and will be trained on FNPA, consistent with standard of care, but the FNPA screening tool will be delayed and phased into care after the intervention period is complete. All PCPs trained but having less than 32 qualifying WCVs will be randomized but excluded from primary outcome analysis. This offers the advantage of concurrently training all PCPs within clinics on standard of care. FNPA has been adopted as standard of care because it facilitates the expected and usual clinical practice of assessing behavioral risks and offering patient-centered preventive care at well child visits. Although all PCPs in clinics will be trained on FNPA, the potential for contamination across arms is low because PCPs in Arm 1 will not have access to the automated


Encircle Protocol Version 1.21 Version Date: 11/29/2022 IRB #: 2020-0207

FNPA for any of their patients until the intervention is complete. PCPs in Arms 2 and 3 will have FNPA all well child visits and be unaware of which children are study participants. There will not be documentation of the Food Care intervention for Arm 3 in the participating child's electronic medical record, thus PCPs will be blind to knowing if they are in Arm 2 or 3 and whether the participant is eligible for Arm 3 Food Care.

Potential child participants will be identified 3 ways: 1) via an electronic medical record data pull performed by a data broker in the Obesity Institute; 2) in the clinic waiting room (pilot); and 3) self-referral. In the electronic health record pathway, the data broker will apply inclusion and exclusion criteria to identify qualifying PCPs and patients that have upcoming well child visits scheduled with a participating PCP. All identified, and potentially eligible participants will be simultaneously sent a recruitment letter, an email (if available), and MyGeisinger message (if available) which provides information regarding the study, participation, how to opt-out, and a study URL and/or QR code to self-refer, and that if they have not contacted the study team, someone will be reaching out by phone to assess interest ( $\geq$ 10 days). The recruitment letter and email for participants will encourage parent proxy enrollment in the patient portal to facilitate communications and scheduling, completion of pre-visit questionnaires in the patient portal (consistent with standard practice), attendance at routine, annual well child visits, and the potential for the intervention to include a health coach and grocery store visit (after the WCV is complete). A reminder email will be sent 3-5 days after the initial email. Participants can completely enroll in the study if they click on/enter the URL/QR code in the email, letter, or portal because all the study enrollment information will available. In the electronic pathway, participants can call or email us with questions they have about the study. After 10 days from sending the letters, the study team will call the participants who did not yet respond electronically and did not opt out. When the potential age-eligible participant does not have history in the electronic health record (e.g., new patient) and the child has an upcoming scheduled well child visit, the study team will call and send an email, letter, and/or MyGeisinger message (if available). When possible, parent/guardians will be provided with 10 days between written or electronic communications and telephone calls; however, calls may occur in a shorter window of time to give the parent/guardian ample opportunity to learn about and participate in the study. This modification acknowledges that patients may be scheduled for a well child visit within a day of calling for an appointment.

Once contacted by phone, the research team will discuss the study with the patient's parent/caregiver, and if the family is interested, obtain informed consent to participate in survey data collection at baseline, 6 months, and 12 months as well as data extraction from their electronic health records. The participant can access the same information by clicking on the URL and/or QR code. Recognizing that participants may experience connectivity difficulties online, the study team will follow-up with participants who start but do not complete the online screening process. E-consent was utilized as the primary consented method for this project until the study team corrected an inefficiency related to the impractability of collecting written consent using a 3-step remote process (call  $\rightarrow$  email  $\rightarrow$  eConsent sign). A waiver of HIPAA authorization was requested to alter the requirement for a written signature and date and replaced by the study team reviewing the consent language with the participant during the screening call and obtaining verbal informed consent. Participants who consent verbally receive a study information sheet and the study team maintains a log of consent authorization. All participants

will have an equal opportunity to participate in this research and will be targeted through multiple attempts using a standard protocol. Telephone calls for recruitment purposes will be performed by Geisinger' Survey Research and Recruitment Center (Call Center) in a secure location housed at the Geisinger Center for Health Research, and accessible only to trained, approved staff.

Novel strategies will be piloted to evaluate the effectiveness of reaching participants as we have been unable to reach more than 40% of participants with electronic/mail/telephone strategies. These strategies will be layered on top of the existing EHR-Identified, electronic/mail/telephone strategies including- in-clinic/in-person, clinical flyer/generic social media, and snowball recruitment. In the pilot in-clinic pathway, potential participants will be screened when they arrive to the clinic. Potential participants will see the study infographic, receive a study flyer, and be screened in the waiting room prior to the well child visit. Enrollment will be contingent on the child meeting inclusion criteria (i.e., BMI will not be known). The study team staff could obtain objectively collected measures from the child's historical electronic health record (before the current WCV) or from the clinic staff. Immediately following the clinical visit, parents of eligible children will complete informed consent and complete baseline questionnaire. Children will be provided with a coloring book and crayons (or other similar materials) to allow the parent time to complete questionnaires. The baseline questionnaire will be broken into 2 parts and evaluated for feasibility of implementation at baseline. For example part A will be brief (5 minutes) to capture parents' attitudes before the visit and allow just enough time for completion before the patient is roomed; part B will be longer (15 minutes). Given that parents may want to leave the clinic immediately following a WCV, especially if a young child is crying after vaccination shots, the study team will follow-up with the parent/guardian to complete consent and baseline data collection following the completed WCV. The in-clinic pilot will occur in less than 5 sites. Workflows will be established with clinical staff to not disrupt care. The in-clinic/in-person recruitment strategy was pilot-tested but discontinued due to low response. In the pilot self-refered pathway, potential participants will respond to to a study flyer posted in the clinic and in social media (e.g., Facebook and/or Instagram). There will be a QR code that sends participants to a self-screening site, similar to the email recruitment strategy. Potential participants and participants will be encouraged to refer a friend using the study flyer. The snowball strategy involves sending a letter and/or email to existing participants asking them to share the opportunity to participate in the study with someone who might be interested. Participants will be provided with a URL, QR code, phone number, email, and study flyer to share with their contact(s). The social media strategy will also utilize patient stories as a potential recruitment method. Results from the pilot efforts will be rapidly evaluated to scale up effective strategies for the remaining study period.

Participant recruitment is based on the Arm of the PCP the child is scheduled with for the upcoming WCV. The patient is recruited up to 6 months prior to the scheduled visit with the intent of being assigned to the treating provider's condition or following a completed WCV. Participant assignment follows PCPs random assignment at the point of scheduling and initial recruitment. The study team expects that most of the participants will see the PCP that they are originally scheduled with or a PCP in the same Arm. However, the study team anticipates that up to 8% of partipants will not receive allocated treatment (i.e., child's WCV is conducted by a PCP in different arm than scheduled) due to absences or unplanned events. In response to this

challenge, the study team will monitor the patient's schedule up to 16-days prior to the WCV. At that point, the study team can modify PRO data collection to the scheduled provider's condition. Two alternate scenarios are planned in the event that the treating provider changes within 16 days of the WCV. First, if a participant is scheduled with an Arm 1 (no PRO) provider but sees an Arm 2/3 provider (PRO view), the participant still has the opportunity to complete PRO in the waiting room because office staff are cued to close open care gaps (PRO) and the participant is reassigned to the treatment provider. Second, if a participant is scheduled with an Arm 2/3 provider (PRO opportunity pre-visit) but sees and Arm 1 provider (no PRO view), then the participant is reassigned to the treating provider. Participants will be retained for intent-to-treat analyses regardless of the PCP Arm at the point of care (WCV). Participants in scenario 1 will be excluded from a per protocol analysis due to limited FNPA exposure and participants in scenario 2 will be excluded from a per protocol analysis due to no opportunity to discuss PRO with the clinical provider. Arm 2 and 3 participants are interchangeable from scheduling assignment through the point of care because the condition is the same through these cases.

Participants in Arm 1 will receive their usual care well child visit with their Arm 1 PCP. They will be asked to complete study questionnaires and return to the same PCP for an annual well child visit (ideally 12 months, 1 day to 17 months, 364 days from baseline well child visit). Participants in Arm 2 and 3 will receive the FNPA screening tool, consistent with standard of care, and asked to complete study questionnaires and return to the same PCP for an annual well child visit (ideally 12 months, 1 day to 17 months, 364 days from baseline well child visit). In December 2020, Geisinger implemented EPIC® standard which included previsit questionnaires, a new feature in the standard licensed software. Changes for participants enrolled in MyGeisinger include the launching of pre-visit surveys at 14 days (rather than 16 days) prior to scheduled visits. The vast majority of study participants are dually enrolled in MyGeisinger and will receive visit reminders via text. Geisinger has requested that EPIC® add functionality for a 'notification tickler' text that will prompt MyGeisinger users to complete standard of care previsit questionnaires (e.g., FNPA) before visits to save time during check-in. Recognizing that the system intends to implement multiple reminders for standard of care questionnaires, the study team requests advance implementation. The rationale: 1) to ensure that a majority of participants will have similar experience to data collection prompts as more than 80% of the sample is yet to be enrolled but the timeline for EPIC® modifications is unknown but likely to occur before study enrollment is complete; and 2) to ensure opportunity for data collection as participants have been refusing to complete pre-visit surveys on Geisinger devices (iPad) in the waiting room, a new phenomena during the COVID pandemic, likely explained by fear of transmission despite clinic staff offering devices and ensuring their cleanliness. Participants in Arms 2 and 3 and who are dually enrolled in MyGeisinger, will receive 3 text message reminders to complete pre-visit questionnaires prior to the well child visit. Sequential reminders are only sent to participants with incomplete questionnaires.

Arm 3 participants will be contacted after the well child visit is complete and offered a referral to the Geisinger Steele Institute Wellness Program (Health Coaches) for the Choose Health LA: Parent Training Program, and a grocery store tour (after the 3<sup>rd</sup> health coach call as learning activities are complementary). The Parent Training Program will be delivered as 6 individual sessions via virtual video (e.g., TEAMS, GoToMeeting, Zoom, Apple FaceTime, Google Duo) or telephone, or video (when participant fails to attend scheduled synchronous

> session), spread throughout a 26-week intervention period. These telephone calls may be recorded to conduct fidelity monitoring in relation to the intervention delivery. The Geisinger Wellness staff will deliver the Choose Health LA curriculum to the study participants as part of their existing roles and responsibilities to advance population health outcomes through outreach and education to patients who screen positive for food insecurity and other social determinants of health. The intent of evaluating the implementation of the Choose Health LA curriculum by Geisinger Wellness is to understand how the curriculum is adapted by staff locally, to inform institutional sustainability, and to inform future implementation and dissemination. The number of Geisinger Wellness staff implementing the curriculum is limited (n=1, 1.0 FTE) and thus, there is no intent to systematically understand how the health coach, per se, affects implementation or outcomes. During the course of the study, other Geisinger staff will be trained to deliver the curriculum if the volume of participants who agree to receive education in Arm 3 exceeds the capacity of existing Wellness 1.0 FTE (or if there is staff turnover). However, there will not likely be more than 3 coaches total in the course of the project, certainly too few to systematically study, and thus will not change the intent of evaluating the implementation of Arm 3.

> Trained study team dietitians may function in the role of the Health Coach in the event of staff shortages; otherwise, the dietitians have no other role on the project. For the purpose of implementation evaluation, Health Coach will be asked to complete questionnaires at baseline, 12- and 24-month follow-up periods. The grocery store tour will be delivered by trained, instore nutritionists across the study region (e.g., Giant Foods, Wegmans, Weis Markets). Grocery store tours are usual practice for in-store nutritionists. To ensure participants are able to receive the grocery store tour trainings, they will be offered both in-person and virtually (utilizing TEAMS, Zoom, etc.) and conducted by the grocery store nutritionists. Patient-preference for delivery (in-person vs. remote or a hybrid) of the Cooking Matters® grocery store tour will be considered to promote participation in the event that social distancing precautions remain in place or participants have transitioned to online grocery ordering. Share Our Strength's Cooking Matters® campaign is increasing efforts to deliver digital content through Zoom, Facebook Live, and YouTube and other platforms to support families with strategies and skills. The study team will collaborate with the in-store nutritionists across the region to utilize newly developed digital content to supplement in-store tour learning activities. Importantly, grocery store nutritionists have also started to transition to virtual care for their customers, thus a transition to digital delivery is consistent with their practice. Participants may receive educational materials by email or postal service mail, per participant preference. In an effort to best track completion of grocery store tours by Arm 3 participants, the study will implement a short Grocery Store Tour questionnaire for participants to complete. This 3-question questionnaire will ask the participant to report if they attended a tour, the grocery chain the tour occurred at, and whether the tour was in-person or online.

The active intervention in Arm 3 will last a total of 6 months with active participant involvement. Participant satisfaction will be collected following the first and last calls with the health coach. Following the 6-month intervention, follow-up measures will be collected at 6 months. For all arms, data will be extracted from the EHR during and following the 12-month period to assess the implementation and impact of the intervention on child BMI.

Participant recruitment is based on the Arm of the PCP the child is scheduled with for the upcoming WCV or completed WCV. Participant assignment follows PCPs random assignment at the point of scheduling and initial recruitment. The study team expects that most of the participants will see the PCP that they are originally scheduled with or a PCP in the same Arm. However, the study team anticipates that participants will be lost when the child does not receive allocated treatment (i.e., child's WCV is conducted by a PCP in different Arm than scheduled) due to absences or unplanned events. Loss of thse participants is accounted for in the sample size for per protocol analyses. However, the primary BMI outcome analysis is an intent- to-treat analyses and will include these children, regardless of the PCP's Arm at the point of care (WCV).

Participants will be reminded to complete study consent, questionnaires, study measures, health coach calls, and grocery store tour via follow-up phone calls, emails, MyGeisinger patient portal, and text messages sent utilizing the internal Geisinger process that is currently leveraged to send appointment reminders to patients. This is an approved platform by ISO.

All data (EHR and patient-self report) will be kept behind the Geisinger firewall on password-protected servers that are only accessible to Geisinger IRB-approved staff. For data shared with PSU, all Geisinger IT/ISO policies regarding secure transportation of patient data will be followed. Data shared outside Geisinger will be stored in a secure location to ensure patient data is protected.

#### **Participant Compensation**

Parents/guardian participants will receive a \$50 check per survey completion at baseline, 6 months, and 12 months for a total of \$150, if the patient completes all 3 surveys, they will receive an additional \$50 for a total of up to \$200. Geisinger providers will not be compensated for completion of study questionnaires. Participating clinics will receive a stipend of \$500-\$1,000 depending on number of qualifying PCPs as those with a higher number may experience greater disruption to workflow with added burden of collecting patient-reported data. Note that all clinics now collect patient-reported data with varied workflows and technology resources (e.g., tablets, kiosks) and this burden is expected to be minimal.

#### **Participant Withdrawal**

Participants who choose to withdraw from the study will not be contacted for further survey data collection. In addition, for participants in Arm 3, if the choice is made to withdraw, they will not receive any further contact from their health coach. Participants may be withdrawn from the study by an investigator if they choose to switch providers or leave Geisinger. All data collected up to the point of withdrawal may be used for analysis purposes.

## **Data Management Procedures and Confidentiality**

Data collected as part of this study will be keep indefinitely for future analysis such as potential follow-up analysis to determine long-term study impacts, and for use in grant planning to pursue additional research-related activities. These data will be stored on stored locally on Geisinger encrypted, password-protected servers behind the Geisinger firewall. Only trained study personnel who adhere to the National Institutes of Health (NIH) policies on the protection

of human subject participants in research, and are approved by the Geisinger IRB, will have access to study data.

Questionnaires will be administered using REDCap, which will also be used to manage and store related data elements (e.g., participant tracking). Data from paper versions of selfadministered questionnaires will be manually entered into an electronic dataset. Double-entry and verification steps will be taken to reduce potential for human error. Electronic questionnaire data will be stored internally on Geisinger's secured network and access to REDCap will be restricted to approved study personnel. Study participant information will not be released to any party without the participant's permission. RedCap access occurs over password-protected channels only accessible via the use of an authenticator. Data is stored locally on Geisinger encrypted, password-protected servers behind the Geisinger firewall.

In the event that data would be transferred outside of Geisinger, it would be done using a secure file transport system maintained by Geisinger IT/ISO. This secure transport method would allow access only to approved IRB study staff with unique usernames and passwords required to access the site.

#### **Data Analysis/ Statistical Considerations**

**Table 2**. Estimated Sample Size per Randomization Arm

| | · | | |
|---|---|---|---|
| Effect size* | e* # Physicians # participan<br>per group Physician | | Total N per group |
| 0.20 | 20 | 32 | 640 |
| 0.20 | 25 | 25 | 625 |
| 0.25 | 20 | 19 | 380 |
| 0.25 | 25 | 15 | 375 |

<sup>\*</sup>Cohen's d: mean difference / SD

#### Sample Size and Power

Our preliminary data comparing the change in BMIz between WCV vs. **PRO WCV** yielded a difference of 0.05 units.<sup>6</sup> This corresponded to an effect size (Cohen's d) of approximately 0.20 of a standard deviation. Additionally, based on our preliminary data and the literature, we estimate the intra-cluster correlation (ICC) to be 0.005 to account for the clustering of participant families within PCP. We recognize that participants may be lost to follow up during the course of the study or that we will not recuit equal number of participant families across all PCPs. Therefore, our sample size calculations further assume a coefficient of variation (COV) equal to 0.25 to account for this potential imbalance. This parameter being greater than 0 (i.e., equal sample size across clusters) increases the required sample size. Lastly, to account for two a priori statistical comparisons in Aim 1 (WCV vs PRO WCV, WCV vs. PRO WCV + Food Care), the significance level is set at 2.5%. Table 2 reports the required sample size for enrollment under the stated assumptions. All calculations assume 80% power and an overall significance level of 5% such that each of the two comparisons will be made at the 2.5% significance level.

The software PASS v15 was used for all calculations, specifically the module for cluster randomized trials for two means. Table 2 reports the required sample size for enrollment under the above stated assumptions (reproduced in this response). We also varied the effect size to additionally include 0.25 and using 20 and 25 PCPs per arm to understand how varying-the


Encircle Protocol Version 1.21 Version Date: 11/29/2022 IRB #: 2020-0207

parameters affected the sample sizes. For example, assuming an effect size of 0.20, ICC of 0.005, COV of 0.25, 80% power, and 0.025 significance level, the study would be required to enroll 28 participant families per PCP per arm for a total of 560 families per arm. However, we further inflated the sample size to account for 7% of participants not receiving allocated treatment (i.e., WCV completed by a PCP in a different Arm than scheduled) and a 10% dropout at 1 year. This yields a sample size of 675 per arm or, with rounding, 33 families per each of 20 PCPs, for a total of 675 per arm (N=2,025 across all three arms).

The study will have 80% power to detect an effect size of 0.20 with 20 PCPs per randomization arm and 33 participant families per PCP, for a total of 2,025 across all three groups in Aim 1. If we are able to obtain more PCPs, then we can reduce the number of families. Also, if the effect size is larger than we observed in our preliminary work,<sup>6</sup> then the study will have > 80%. It is recognized that to assess for mediation and moderation that a larger sample size is required and thus, we do not expect to have a large power to detect these effects. Thus, Aim 2 results will be descriptive in nature. Given that multiple recruitment strategies are simultaneously in place, and the rate of enrollment is about 10 participants/week when 95% of the targeted sample has been achieved, the study has a buffer of 15 additional participants who may be in latter stages of recruitment when the sample is achieved. In other words, up to 2040 participants may be enrolled.

#### **Outcomes**

The primary child-level outcome is the 1-year difference in change in BMIz between study arms using World Health Organization growth reference standards. BMI values will be obtained from Geisinger clinical care visits, documented in the EHR. Values obtained at well child visits (preferred), clinical visits, or self-report during the study period, ideally 12 months, 1 day apart will be utilized but values from baseline WCV to 9 to 18 month follow-up may be used to assess the primary outcome. This primary outcome is chosen because it reflects the difference in the effectiveness of each intervention versus standard of care in preventing obesity among a highrisk population of preschool-aged children. The difference in the difference between groups is chosen because the intervention is randomized at the PCP and not the patient-level. Parent selfreport of child weight and height is added to supplement primary outcome data given unprecedented changes in pediatric care secondary to the pandemic. Specifically, the availability of WCVs has decreased due to staff turnovers yet the demand has decreased as families delay or forgo preventive care. To optimize follow-up height and weight data collection, parents of children without a clinical BMI at about 1-year post-baseline WCV, will be encouraged to complete the child's follow-up WCV, per clinical schedule, or to visit the clinic for height and weight measures. Among this subset of the study population (implemented in September 2022), parent self-reported data about child's height and weight will be collected before the WCV or clinic visit. 153-156 Parents will be asked whether the self-reported data are estimates or measured at home. 153-156 Among a smaller subset, the self-reported data will be compared with objective height and weight collected in usual clinical care. Concordance between the parent self-report and clinical measures will be evaluated for validation of self-reported data. If the variation among self-report with objective clinical measures is acceptable, self-reported data may be used as follow-up measures. To determine if the variation is acceptable, variation will be compared to the literature to inform analytical strategies for using supplmental parent-reported data in the absence of clinical measures. 153-156 The use of self-reported measures is anticipated for studies

> conducted during the pandemic and will likely be found in emerging and current literature. 157 While many adiposity outcomes could be used, this outcome will facilitate interpretation of the relevance of the findings among PCPs, health care administrators, policy makers, and researchers who pursue future systematic reviews of delivery care models to prevent childhood obesity. Nonetheless, BMIz can be too restrictive to evaluate success and may not be meaningful to parents or clinicians. 122 Therefore, we will also evaluate the proportion of children overweight and obese at 1-year follow-up per CDC guidance and definitions (https://www.cdc.gov/obesity/childhood/defining.html), difference in raw BMI and difference in BMI50 between study arms, and BMIz extended. 158-160 Patient stakeholders to the project (Patient Advisory Council on Obesity, PACO) identified meaningful secondary outcomes and PCP's identified mediating pathways to inform steps that parents and PCPs can take together to prevent obesity. Specifically, findings will help to inform parents of what they can realistically expect for their children if they pursue standard of care WCV, complete the PRO risk assessment and engage in discussion with their child's PCP, or take these steps and participate in a community-based nutrition program. PCPs would understand benefit of utilizing FNPA, training, and intentionally engaging parents in counseling on childhood obesity prevention.

#### **Analytic Plan**

During the start-up of the study we will develop a formal Data Management Plan to document how data will be collected, organized, stored, as well as a statistical analysis plan. Descriptive statistics will include evaluation of all data for underlying distribution and summary statistics, using means with standard deviations and medians with interquartile range for continuous variables, and frequency with percentages for categorical variables. The data will be summarized for all patients enrolled and will be stratified by randomization arm and study time point. We will assess the quality of data, evaluating outliers and patterns of missing data using graphs such as histograms and stem-and-leaf plots. Bi-variate analyses will be used to assess differences in patients (e.g., parent BMI, child biological sex, baseline BMI) between randomization arms. Since it is not recommended to perform inferential statistics to assess balance of baseline participant, family, community, and physician factors in a randomized study, we will use standardized differences. Any standardized difference > 0.10 will be considered unbalanced and, thus, a potential confounding variable. We will also follow the CONSORT extension to cluster randomized trials when reporting results.

As data is collected from participants as part of this research study, in an effort to facilitate additional analyses, the Geisinger study team plans to share a de-identified data set with PSU. This data set will be shared utilized Geisinger IT-approved methodologies (Secure Transport, e-secure, etc.) to ensure that patient data is protected. These data will be stored at PSU in a secure network location that is only accessible to PSU study staff. These analyses will assist in exploring additional study research questions that may arise.

**Aim 1.** The primary outcome variable is change in BMIz at 12 months. BMIz is the most widely used obesity-related outcome per systematic review and thus was chosen for comparability with prior literature. 11,105 The primary analysis will follow the "intention-to-treat" principal. That is, all participants enrolled will be analyzed according to their group assignment at the point of care (WCV) regardless of intervention received and compliance. Analyses will

> take into account the clustered nature of the study design. To test the Aim 1 hypothesis that participants will have a lower change in BMIz (and secondarily, changes in BMI, BMI50, BMIz extended) in Arms 2 and 3, as compared to Arm 1, mixed linear models 106,107 with restricted maximum likelihood estimation will be fit. The models will include a random effect for PCPs and will be assumed to follow a Gaussian distribution. These analyses will adjust for the stratification factors used in the randomization scheme and any baseline variables found to vary across intervention arms as identified above. Contrast statements will be written as functions of the estimated regression coefficients to estimate the effect of the interventions compared to standard WCV using a two-sided alpha of 0.025 to account for multiple testing. Model assumptions will be examined (e.g., QQ plots to assess normally distributed residuals) and of the underlying Gaussian random effect distribution. Secondary analyses will estimate the effectiveness of the interventions on the percent of children overweight and obese (> 85 percentile of BMI and > 95 percentile of BMI) at 12 months. A similar strategy will be employed using a generalized linear mixed model assuming a binomial distribution for the outcomes. These models will treat the binary outcomes as measured from the 12-month visit. Analysis of secondary outcomes in Aims 1b and 1c (involvement in preventive care, parent and home factors) will follow the same strategy as described above. Due to lagging enrollment, the study modified data collection for secondary outcome in specific aim 1b- involvement in preventive care- just after 50% enrollment was reached. The timing of this outcome measure was changed from pre-visit only to pre- or -post visit to allow for families to enroll and complete baseline data collection after a completed WCV. As there are complementary analysis methods for cluster randomized trials, we will also fit Bayesian random effect models 108-110 for continuous and binary outcomes. Each model will use an inverse gamma prior for the cluster random effect variance parameter. 111 We will note any differences in the effect estimates across methods.

> **Aim 2.** The primary outcome variable is the same as in Aim 1, change in BMIz at 12 months. Aim 2 involves the assessment of mediating and moderating effects of PCP, parental and child behaviors (see list of variables in **Appendix B**). For a variable to be considered a mediator it must be associated with and in the casual pathway between the intervention and outcome. Therefore, we will first fit mixed linear models to each hypothesized mediator as dependent variables following the approach described in Aim 1. We will then fit similar models with BMIz as the outcome and each potential mediator as independent variable. Any variable found to be associated with intervention and BMIz will be considered a potential mediator variable. Our list of candidate mediator variables is measured at both the subject (parent and child) and cluster levels (PCP). To appropriately fit models with mediation at different levels we will rewrite the mixed models of Aim 1 as multilevel structure equation models (MSEM)<sup>112</sup> to include the variables in the analysis. Results will be expressed as total, direct, and indirect effects as estimated from the model. Moderation will be assessed using the MSEM framework. 113 In Aim 1, we will also fit complementary Bayesian models to assess robustness of effect estimates. Aim 2 outcomes may be evaluated using secondary outcomes including raw BMI, BMI50, and BMIz extended.

**Missing Data Considerations.** We will minimize missing data by querying the EHR for anticipated and scheduled 1-year follow-up WCVs, sending reminders to each participant to schedule and attend appointment, and reminding participants of 1-year follow-up study questionnaires. Missing data, however, are inevitable in a longitudinal study due to dropout and

> nonresponse to study questionnaire items. We anticipate that no more than 7% of randomized subjects will not receive allocated treatment and 10% of randomized subjects will fail to complete the study; 63,90,115 but reasons for loss at point of WCV care and dropout will be documented. Before proceeding with primary analyses, we will characterize patterns of missingness using exploratory analyses to provide insights into how to handle the missing data. Participants with missing data will be compared to participants with complete data to ensure there are no differences. Depending on the amount of missing data, we will use a non-parametric missing data imputation method based on random forests. 116 This method has been shown to perform as well as or better than more traditional methods of imputation, and it has the advantage of imputing both continuous and categorical data. By using random forests, we can capture non-linear relationships and interactions present in the dataset that may otherwise be missed when using a different method. At least 5 complete datasets will be created and combined using the methods of Rubin.<sup>117</sup>

Heterogeneity of treatment effect (HTE). HTE analyses are incorporated into Aim 2 when examining moderator effects. Additional sub-group analyses will be performed by child sex (males, females) and baseline BMI weight category (overweight, obese). These sub-group analyses will employ the same models as described in Aim 2.

Aim 3. The RE-AIM framework<sup>29</sup> will be used to evaluate the interventions' reach to the target population and subgroups (e.g., by provider type, those with food insecurity and hunger), comparative effectiveness, adoption by PCPs, implementation fidelity and barriers, and maintenance of intervention components over time, so as to inform translation of this study into practice.

#### **EXPECTED RISKS/ BENEFITS**

#### **Potential Risks**

The greatest potential risk to participants in this research is a loss of confidentiality. To minimize the risk of loss of confidentiality, all data collected as part of this study will be stored on the Geisinger password-protected network only accessible to IRB-approved study staff. Participants will also be assigned a unique study ID for data collection. In the event that any data would be shared outside of Geisinger, it would be done using an IT-approved secure transport method to ensure data security is maintained.

#### **Benefits**

By participating in this study, participants may experience direct benefits from familycentered care for early childhood obesity prevention. Their participation may help researchers and Geisinger develop ways to improve the care of pediatric patients. Although individual study participants will not benefit, we believe the minimal risks they face by participating are reasonable give the potential benefit future patients may receive related to pediatric obesity prevention.

#### **BIBLIOGRAPHY**

1. Glass TA, McAtee MJ. Behavioral science at the crossroads in public health: extending horizons, envisioning the future. *Soc Sci Med.* 2006;62(7):1650-71.

- 2. Geserick M, Vogel M, Gausche R, Lipek T, Spielau U, Keller E, Pfäffle R, Kiess W, Körner A. Acceleration of BMI in early childhood and risk of sustained obesity. *N Engl J Med*. 2018;379(14):1303-12.
- 3. Nader PR, O'Brien M, Houts R, Bradley R, Belsky J, Crosnoe R, Friedman S, Mei Z, Susman EJ. Identifying risk for obesity in early childhood. *Pediatrics*. 2006;118(3):e594-601.
- 4. Bailey-Davis L, Kling SM, Cochran WJ, Hassink S, Hess L, Franceschelli Hosterman J, Lutcher S, Marini M, Mowery J, Paul IM, Savage JS. Integrating and coordinating care between the Women, Infants, and Children Program and pediatricians to improve patient-centered preventive care for healthy growth. *Transl Behav Med*. 2018;8(6):944-52.
- 5. American Academy of Pediatrics. Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999–2016. *Pediatrics*. 2018; 141 (3): e20173459. *Pediatrics*. 2018 Sep 1;142(3):e20181916.
- 6. Bailey-Davis L, Kling SM, Wood GC, Cochran WJ, Mowery JW, Savage JS, Stametz RA, Welk GJ. Feasibility of enhancing well child visits with family nutrition and physical activity risk assessment on body mass index. *Obesity Science & Practice*. 2019 Apr 24;5(3):220-230. doi: 10.1002/osp4.339. eCollection 2019 Jun. PMID:31275595
- 7. Taveras EM, Marshall R, Sharifi M, Avalon E, Fiechtner L, Horan C, Gerber MW, Orav EJ, Price SN, Sequist T, Slater D. Comparative effectiveness of clinical-community childhood obesity interventions: a randomized clinical trial. *JAMA Pediatrics*. 2017;171(8):e171325.
- 8. Slusser W, Frankel F, Robison K, Fischer H, Cumberland WG, Neumann C. Pediatric overweight prevention through a parent training program for 2–4 year old Latino children. *Child Obes*. 2012 Feb;8(1):52-9.
- 9. Barlow SE. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. *Pediatrics*. 2007;120(Suppl 4):S164-92.
- 10. Daniels SR, Hassink SG. The role of the pediatrician in primary prevention of obesity. *Pediatrics*. 2015;136(1):e275-92.
- 11. Wang Y, Cai L, Wu Y, Wilson RF, Weston C, Fawole O, Bleich SN, Cheskin LJ, Showell NN, Lau BD, Chiu DT. What childhood obesity prevention programmes work? A systematic review and meta-analysis. *Obes Rev.* 2015 Jul;16(7):547-65.
- 12. Ogden CL, Fryar CD, Hales CM, Carroll MD, Aoki Y, Freedman DS. Differences in Obesity Prevalence by Demographics and Urbanization in US Children and Adolescents, 2013-2016. *JAMA*. 2018;319(23):2410-8.
- 13. Befort CA, Nazir N, Perri MG. Prevalence of obesity among adults from rural and urban areas of the United States: Findings from NHANES (2005-2008). *J Rural Health*. 2012; 28:392-397.
- 14. Bailey-Davis L, Horst M, Hillemeier MM, Lauter A. Obesity disparities among elementary-aged children: Data from school-based BMI surveillance. *Pediatrics*. 2012;130(6): 1102-1109.

15. Johnson JA, Johnson AM. Urban-rural differences in childhood and adolescent obesity in the United States: a systematic review and meta-analysis. *Child Obes*. 2015;11(3):233-41.

- 16. Savage JS, Kling SM, Cook A, Hess L, Lutcher S, Marini M, Mowery J, Hayward S, Hassink S, Hosterman JF, Paul IM. A patient-centered, coordinated care approach delivered by community and pediatric primary care providers to promote responsive parenting: pragmatic randomized clinical trial rationale and protocol. *BMC Pediatr*. 2018;18(1):293.
- 17. Adler NE, Stead WW. Patients in context—EHR capture of social and behavioral determinants of health. *N Engl J Med*. 2015;372(8):698-701.
- 18. Glasgow RE, Kaplan RM, Ockene JK, Fisher EB, Emmons KM. Patient-reported measures of psychosocial issues and health behavior should be added to electronic health records. *Health Aff (Millwood)*. 2012;31(3):497-504.
- 19. Christison A, Daley B, Asche C, et al. Pairing motivational interviewing with a nutrition and physical activity assessment and counseling tool in pediatric clinical practice: A pilot study. *Child Obes*. 2014;10:432-441.
- 20. JaKa MM, Seburg EM, French SA, Wolfson J, Jeffery RW, Levy RL, Langer SL, Sherwood NE. Parent Choice in a Pediatric Obesity Prevention Intervention. *Health Behav Policy Rev.* 2017;4(4):357-66.
- 21. Dietz WH, Solomon LS, Pronk N, et al. An integrated framework for the prevention and treatment of obesity and its related chronic diseases. *Health Aff (Millwood)*. 2015;34(9):1456-63.
- 22. Dietz WH, Belay B, Bradley D, Kahan S, Muth ND, Sanchez E, Solomon L. A model framework that integrates community and clinical systems for the prevention and management of obesity and other chronic diseases. National Academy of Medicine; 2017 Jan 13; Washington, DC.
- 23. Pooler JA, Morgan RE, Wong K, Wilkin MK, Blitstein JL. Cooking Matters for Adults improves food resource management skills and self-confidence among low-income participants. *J Nutr Educ Behav*. 2017;49(7):545-53.
- 24. Mabli J, Ohls J, Dragoset L, Castner L, Santos B. Measuring the effect of Supplemental Nutrition Assistance Program (SNAP) participation on food security. Mathematica Policy Research. 2013 Aug 30.
- 25. Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. *Appetite*. 2001;36(3):201-10.
- 26. Ventura AK, Birch LL. Does parenting affect children's eating and weight status?. *Int J Behav Nutr Phys Act.* 2008;5(1):15.
- 27. Nau C, Schwartz BS, Bandeen-Roche K, Liu A, Pollak J, Hirsch A, Bailey-Davis L, Glass TA. Community socioeconomic deprivation and obesity trajectories in children using electronic health records. *Obesity (Silver Spring)*. 2015 Jan;23(1):207-12.
- 28. Ohri-Vachaspati P, DeLia D, DeWeese RS, Crespo NC, Todd M, Yedidia MJ. The relative contribution of layers of the Social Ecological Model to childhood obesity. *Public Health Nutr.* 2015;18(11):2055-66.

- 29. Klesges LM, Estabrooks PA, Dzewaltowski DA, Bull SS, Glasgow RE. Beginning with the application in mind: designing and planning health behavior change interventions to enhance dissemination. *Ann Behav Med.* 2005;29(2):66-75.
- 30. Hales CM, Fryar CD, Carroll MD, Freedman DS, Ogden CL. Trends in obesity and severe obesity prevalence in US youth and adults by sex and age, 2007-2008 to 2015-2016. *JAMA*. 2018;319(16):1723-5.
- 31. Tamayo T, Herder C, Rathmann W. Impact of early psychosocial factors (childhood socioeconomic factors and adversities) on future risk of type 2 diabetes, metabolic disturbances and obesity: a systematic review. *BMC Public Health*. 2010;10(1):525.
- 32. Friedemann C, Heneghan C, Mahtani K, Thompson M, Perera R, Ward AM. Cardiovascular disease risk in healthy children and its association with body mass index: systematic review and meta-analysis. *BMJ*. 2012;345:e4759.
- 33. Skinner AC, Perrin EM, Moss LA, Skelton JA. Cardiometabolic risks and severity of obesity in children and young adults. *N Engl J Med*. 2015;373(14):1307-17.
- 34. Bocca G, Ongering EC, Stolk RP, Sauer PJ. Insulin resistance and cardiovascular risk factors in 3-to 5-year-old overweight or obese children. *Horm Res Paediatr*. 2013;80(3):201-6.
- 35. May AL, Kuklina EV, Yoon PW. Prevalence of cardiovascular disease risk factors among US adolescents, 1999-2008. *Pediatrics*. 2012;129(6):1035.
- 36. Egan KB, Ettinger AS, Bracken MB. Childhood body mass index and subsequent physician-diagnosed asthma: a systematic review and meta-analysis of prospective cohort studies. *BMC Pediatrics*. 2013;13(1):121.
- 37. Bell LM, Byrne S, Thompson A, Ratnam N, Blair E, Bulsara M, Jones TW, Davis EA. Increasing body mass index z-score is continuously associated with complications of overweight in children, even in the healthy weight range. *J Clin Endocrinol Metab*. 2006;92(2):517-22.
- 38. Griffiths LJ, Parsons TJ, Hill AJ. Self-esteem and quality of life in obese children and adolescents: a systematic review. *Int J Pediatr Obes*. 2010;5(4):282-304.
- 39. Simmonds M, Burch J, Llewellyn A, Griffiths C, Yang H, Owen C, Duffy S, Woolacott N. The use of measures of obesity in childhood for predicting obesity and the development of obesity-related diseases in adulthood: a systematic review and meta-analysis. *Health Technol Assess.* 2015;19(43):1-336.
- Ward ZJ, Long MW, Resch SC, Giles CM, Cradock AL, Gortmaker SL. Simulation of growth trajectories of childhood obesity into adulthood. N Engl J Med. 2017;377(22):2145-53.
- 41. Blake-Lamb TL, Locks LM, Perkins ME, Baidal JA, Cheng ER, Taveras EM. Interventions for childhood obesity in the first 1,000 days a systematic review. American journal of preventive medicine. 2016 Jun 1;50(6):780-9.
- 42. Baidal JA, Locks LM, Cheng ER, Blake-Lamb TL, Perkins ME, Taveras EM. Risk factors for childhood obesity in the first 1,000 days: a systematic review. American journal of preventive medicine. 2016 Jun 1;50(6):761-79.
- 43. Ash T, Agaronov A, Aftosmes-Tobio A, Davison KK. Family-based childhood obesity prevention interventions: a systematic review and quantitative content analysis. *Int J Behav Nutr Phys Act.* 2017;14(1):113.

- 44. Huang TT, Borowski LA, Liu B, Galuska DA, Ballard-Barbash R, Yanovski SZ, Olster DH, Atienza AA, Smith AW. Pediatricians' and family physicians' weight-related care of children in the US. *Am J Prev Med*. 2011;41(1):24-32.
- 45. Te Morenga L, Mallard S, Mann J. Dietary sugars and body weight: systematic review and meta-analyses of randomised controlled trials and cohort studies. *BMJ*. 2013;346:e7492.
- 46. Cox R, Skouteris H, Rutherford L, Fuller-Tyszkiewicz M, Dell D, Hardy LL. Television viewing, television content, food intake, physical activity and body mass index: a cross-sectional study of preschool children aged 2-6 years. *Health Promot J Austr*. 2012;23(1):58-62.
- 47. Tremblay MS, LeBlanc AG, Kho ME, Saunders TJ, Larouche R, Colley RC, Goldfield G, Gorber SC. Systematic review of sedentary behaviour and health indicators in schoolaged children and youth. *Int J Behav Nutr Phys Act*. 2011;8(1):98.
- 48. Fatima Y, Doi SA, Mamun AA. Longitudinal impact of sleep on overweight and obesity in children and adolescents: a systematic review and bias-adjusted meta-analysis. *Obes Rev.* 2015;16(2):137-49.
- 49. Perez-Escamilla R, Segura-Perez S, Lott M. on behalf of the RWJF HER Expert Panel on Best Practices for Promoting Healthy Nutrition, Feeding Patterns, and Weight Status for Infants and Toddlers from Birth to 24 Months. Feeding Guidelines for Infants and Young Toddlers: A Responsive Parenting Approach. 2017; Durham, NC.
- 50. Ihmels M, Welk G, Eisenmann J, Nusser S. Development and preliminary validation of a family nutrition and physical activity (FNPA) screening tool. *Int J Behav Nutr Phys Act*. 2009;6.
- 51. Ihmels M, Welk G, Eisenmann J, Nusser S, Myers E. Prediction of BMI change in young children with the family nutrition and physical activity (FNPA) screening tool. *Ann Behav Med.* 2009:38:60-68.
- 52. Peyer KL, Welk GJ. Construct validity of an obesity risk screening tool in two age groups. *Int J Environ Res Public Health*. 2017;14(4):10.3390/ijerph14040419. doi: E419.
- 53. Yee K, Eisenmann J, Calson J, Pfeiffer K. Association between the family nutrition and physical activity screening tool and cardiovascular disease risk factors in 10-year old children. *Int J Pediatr Obes.* 2011;6:314-320.
- 54. Yee KE, Pfeiffer KA, Turek K, et al. Association of the family nutrition and physical activity screening tool with weight status, percent body fat, and acanthosis nigricans in children from a low socioeconomic, urban community. *Ethn Dis.* 2015;25(4):399-404. doi: 10.18865/ed.25.4.399.
- 55. Tucker JM, Howard K, Guseman EH, Yee KE, Saturley H, Eisenmann JC. Association between the Family Nutrition and Physical Activity Screening Tool and obesity severity in youth referred to weight management. *Obes Res Clin Pract*. 2017;11(3):268-75.
- 56. Bleich SN, Segal J, Wu Y, Wilson R, Wang Y. Systematic review of community-based childhood obesity prevention studies. *Pediatrics*. 2013;132(1):e201-10.
- 57. Waters E, de Silva-Sanigorski A, Burford BJ, Brown T, Campbell KJ, Gao Y, Armstrong R, Prosser L, Summerbell CD. Interventions for preventing obesity in children. *Cochrane Database Syst Rev.* 2011(12).

58. Stice E, Shaw H, Marti CN. A meta-analytic review of obesity prevention programs for children and adolescents: the skinny on interventions that work. *Psychol Bull*. 2006;132(5):667.

- 59. Poulsen MN, Bailey-Davis L, Pollak J, Hirsch AG, Schwartz BS. Household Food Insecurity and Home Food Availability in Relation to Youth Diet, Body Mass Index, and Adiposity. *J Acad Nutr Diet*. 2019 Mar 8.
- 60. Frongillo EA, Bernal J. Understanding the coexistence of food insecurity and obesity. *Current Pediatrics Reports*. 2014;2:284-290.
- 61. Eisenmann JC, Gundersen C, Lohman BJ, Garasky S, Stewart SD. Is food insecurity related to overweight and obesity in children and adolescents? A summary of studies, 1995-2009. *Obes Rev.* 2011;12(5):e73-83.
- 62. Franklin B, Jones A, Love D, Puckett S, Macklin J, White-Means S. Exploring mediators of food insecurity and obesity: a review of recent literature. *J Community Health*. 2012;37(1):253-264.
- 63. Barkin SL, Heerman WJ, Sommer EC, Martin NC, Buchowski MS, Schlundt D, Po'e EK, Burgess LE, Escarfuller J, Pratt C, Truesdale KP. Effect of a behavioral intervention for underserved preschool-age children on change in body mass index: a randomized clinical trial. *JAMA*. 2018 Aug 7;320(5):450-60.
- 64. Hager ER, Quigg AM, Black MM, Coleman SM, Heeren T, Rose-Jacobs R, Cook JT, de Cuba SA, Casey PH, Chilton M, Cutts DB. Development and validity of a 2-item screen to identify families at risk for food insecurity. *Pediatrics*. 2010;126(1):e26-32.
- 65. Palakshappa D, Vasan A, Khan S, Seifu L, Feudtner C, Fiks AG. Clinicians' perceptions of screening for food insecurity in suburban pediatric practice. *Pediatrics*. 2017;140(1):e20170319.
- 66. Higginbotham K, Crutcher TD, Karp SM. Screening for Social Determinants of Health at Well-Child Appointments: A Quality Improvement Project. *Nurs Clin North Am*. 2019;54(1):141-8.
- 67. Fiechtner L, Puente GC, Sharifi M, Block JP, Price S, Marshall R, Blossom J, Gerber MW, Taveras EM. A Community Resource Map to Support Clinical-Community Linkages in a Randomized Controlled Trial of Childhood Obesity, Eastern Massachusetts, 2014-2016. *Prev Chronic Dis.* 2017;14:E53.
- 68. Evidence for Action. What is a Culture or Health? Accessed online May 22, 2017 at: <a href="http://www.evidenceforaction.org/what-culture-health">http://www.evidenceforaction.org/what-culture-health</a>.
- 69. Glasgow RE, Tracy Orleans C, Wagner EH, Curry SJ, Solberg LI. Does the chronic care model serve also as a template for improving prevention?. *Milbank Q*. 2001;79(4):579-612.
- 70. Martin LT, Plough A, Carman KG, Leviton L, Bogdan O, Miller CE. Strengthening Integration Of Health Services And Systems. *Health Aff (Millwood)*. 2016;35(11):1976-1981.
- 71. Siegel RM, Haemer M, Kharofa RY, Christison AL, Hampl SE, Tinajero-Deck L, Lockhart MK, Reich S, Pont SJ, Stratbucker W, Robinson TN. Community Healthcare and Technology to Enhance Communication in Pediatric Obesity Care: Expert Exchange Workgroup's Views. *Childhood Obesity*. 2018 Jun 7.

72. SNAP-Ed Plan Guidance and Templates. United States Department of Agriculture. Accessed online January 17, 2019 at: https://snaped.fns.usda.gov/sites/default/files/documents/Section1.pdf.

- 73. Center for Childhood Obesity Research. The Pennsylvania State University. Accessed online January 17, 2019 at: https://hhd.psu.edu/ccor.
- 74. Schlechter CR, Rosenkranz RR, Guagliano JM, Dzewaltowski DA. A systematic review of children's dietary interventions with parents as change agents: Application of the RE-AIM framework. *Prev Med.* 2016;91:233-43.
- 75. Davison KK, Birch LL. Childhood overweight: a contextual model and recommendations for future research. *Obes Rev.* 2001;2(3):159-71.
- 76. Lobstein T, Baur L, Uauy R. Obesity in children and young people: a crisis in public health. *Obes Rev.* 2004;5:4-85.
- 77. Ajzen, Icek. The theory of planned behaviour: reactions and reflections. *Psychol Health*. 2011; 26(9): 1113-1127.
- 78. Andrews KR, Silk KS, Eneli IU. Parents as health promoters: A theory of planned behavior perspective on the prevention of childhood obesity. *J Health Commun*. 2010;15(1):95-107.
- 79. Frankfurter C, Cunningham C, Morrison KM, Rimas H, Bailey K. Understanding academic clinicians' intent to treat pediatric obesity. *World J Clin Pediatr*. 2017;6(1):60.
- 80. Pellecchia M, Beidas RS, Marcus SC, Fishman J, Kimberly JR, Cannuscio CC, Reisinger EM, Rump K, Mandell DS. Study protocol: implementation of a computer-assisted intervention for autism in schools: a hybrid type II cluster randomized effectiveness-implementation trial. *Implement Sci.* 2016;11(1):154.
- 81. Williams NJ. Assessing mental health clinicians' intentions to adopt evidence-based treatments: reliability and validity testing of the evidence-based treatment intentions scale. *Implement Sci.* 2015;11(1):60.
- 82. AAP Recommendations for Preventive Pediatric Health Care. Accessed online April 22, 2019 at: (https://www.aap.org/en-us/documents/periodicity\_schedule.pdf
- 83. Saviñon C, Taylor JS, Canty-Mitchell J, Blood-Siegfried J. Childhood obesity: can electronic medical records customized with clinical practice guidelines improve screening and diagnosis?. *J Am Acad Nurse Pract*. 2012;24(8):463-71.
- 84. Choose Health LA. Accessed online April 22, 2019 at: <a href="http://goodfood.ucla.edu/k-12-school-food-resource-toolkit/service/choose-health-la-parent-training-curriculum">http://goodfood.ucla.edu/k-12-school-food-resource-toolkit/service/choose-health-la-parent-training-curriculum</a>.
- 85. Cooking Matters EXTRA for Parents of Preschoolers. SNAP-Ed Toolkit: Obesity Prevention Interventions and Evaluation Framework. Accessed online January 17, 2019 at: <a href="https://snapedtoolkit.org/interventions/programs/cooking-matters/">https://snapedtoolkit.org/interventions/programs/cooking-matters/</a>.PA Tracks, 2018 Statewide Needs Assessment. Accessed online April 22, 2019 at: <a href="https://sites.psu.edu/fy18pasnapedrfp/files/2017/01/FY18\_RFP\_StatewideNeedsAssessment-lirz59m.pdf">https://sites.psu.edu/fy18pasnapedrfp/files/2017/01/FY18\_RFP\_StatewideNeedsAssessment-lirz59m.pdf</a>.
- 86. Taveras EM, Marshall R, Sharifi M, Avalon E, Fiechtner L, Horan C, Orav J, Price SN, Sequist T, Slater D. Connect for Health: Design of a clinical-community childhood obesity intervention testing best practices of positive outliers. *Contemporary Clinical Trials*. 2015;45(Pt B):287-295.
- 87. Chang AR, Bailey-Davis L, Hetherington V, Ziegler A, Yule C, Kwiecen S, Graboski E, Melough MM, Collins C, Anderson C. Remote Dietary Counseling Using Smartphone

- Applications in Patients With Stages 1-3a Chronic Kidney Disease: A Mixed Methods Feasibility Study. Journal of Renal Nutrition. 2019 May 8.
- 88. Wood C, Bailey-Davis L, Mowery J, Seiler C, Cook A, Cunningham K, Naylor A, Jamieson S, Rolston D, Still C. Communicating Personalized Diabetes Risk with Options for Weight Management: Recruitment, Enrollment, and Outcomes. Abstracts from the 25<sup>th</sup> annual Health Care Systems Research Network. *J Patient Cent Res Rev*, 2019;6(1):52-126.
- 89. French SA, Sherwood NE, Veblen-Mortenson S, Crain AL, JaKa MM, Mitchell NR, Hotop AM, Berge JM, Kunin Batson AS, Truesdale K, Stevens J. Multicomponent Obesity Prevention Intervention in Low-Income Preschoolers: Primary and Subgroup Analyses of the NET-Works Randomized Clinical Trial, 2012–2017. *Am J Public Health*. 2018;108(12):1695-706.
- 90. Grossman DC, Bibbins-Domingo K, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Epling JW, Kemper AR, Krist AH, Kurth AE, Landefeld CS. Screening for obesity in children and adolescents: US Preventive Services Task Force recommendation statement. JAMA. 2017 Jun 20;317(23):2417-26.
- 91. Pinard CA, Uvena LM, Quam JB, Smith TM, Yaroch AL. Development and testing of a revised cooking matters for adults survey. *Am J Health Behav*. 2015;39(6):866-73.
- 92. Kaiser L, Chaidez V, Algert S, Horowitz M, Martin A, Mendoza C, Neelon M, Ginsburg DC. Food resource management education with SNAP participation improves food security. *J Nutr Educ Behav.* 2015;47(4):374-8.
- 93. Rivera RL, Maulding MK, Abbott AR, Craig BA, Eicher-Miller HA. SNAP-Ed (Supplemental Nutrition Assistance Program–Education) Increases Long-Term Food Security among Indiana Households with Children in a Randomized Controlled Study–4. *J Nutr.* 2016;146(11):2375-82.
- 94. USDA Nutrition Education and Obesity Prevention Program. FY2020 SNAP-Ed Plan Guidance. 2019. <a href="https://snaped.fns.usda.gov/sites/default/files/documents/SNAP-Ed%20Plan%20Guidance%20FY%202020%20Complete.pdf">https://snaped.fns.usda.gov/sites/default/files/documents/SNAP-Ed%20Plan%20Guidance%20FY%202020%20Complete.pdf</a>. Accessed online December 24, 2019.
- 95. Hess A, Passaretti M, & Coolbaugh S. Fresh Food Farmacy. *American Journal of Health Promotion*. 2019; *33*(5),830–832.
- 96. Talbot JA, Burgess AR, Thayer D, Parenteau L, Paluso N, Coburn AF. Patterns of telehealth use among rural Medicaid beneficiaries. The Journal of Rural Health. 2019 Jun;35(3):298-307.
- 97. Klitzman P, Armstrong B, Janicke DM. Distance as a predictor of treatment attendance in a family based pediatric weight management program in rural areas. The Journal of rural health. 2015 Jan;31(1):19-26.
- 98. Ballard DW, Vemula R, Chettipally UK, Kene MV, Mark DG, Elms AK, Lin JS, Reed ME, Huang J, Rauchwerger AS, Vinson DR. Optimizing clinical decision support in the electronic health record. *Appl Clin Inform*. 2016;7(03):883-98.
- 99. Ali SM, Giordano R, Lakhani S, Walker DM. A review of randomized controlled trials of medical record powered clinical decision support system to improve quality of diabetes care. *Int J Med Inform.* 2016;87:91-100.
- 100. Kling, SMR, Harris HA, Hess LB, Lutcher S, Marini M, Mowery JW, Savage JS, Bailey-Davis L. Integrated framework for early obesity prevention engages parents,

- pediatric clinical care, and community nutrition services as a strategy to advance population health. (under review).
- 101. Totten AM, Womack DM, Eden KB, McDonagh MS, Griffin JC, Grusing S, Hersh WR. Telehealth: Mapping the Evidence for Patient Outcomes from Systematic Reviews. Technical Brief No 25. (Prepared by the Pacific Northwest Evidence-based Practice Center under Contract No. 290-2015-00009-I.) AHRQ Publication No. 16-EHC034-EF. Rockville, MD: Agency for Healthcare Research and Quality; June 2016. <a href="https://www.effectivehealthcare.ahrq.gov/reports/final.cfm">www.effectivehealthcare.ahrq.gov/reports/final.cfm</a>. Accessed online December 24, 2019.
- 102. Austin PC, Balance Diagnostics for Comparing the Distribution of Baseline Covariates between Treatment Groups in Propensity-Score Matched Samples. *Stat Med*. 2009;28(25):2083-3107.
- 103. Campbell MK, Piaggio G, Elbourne DR, Altman DG; for the CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. *BMJ*. 2012;345:e5661.
- 104. Cole TJ, Faith MS, Pietrobelli A, Heo M. What is the best measure of adiposity change in growing children: BMI, BMI%, BMI z-score or BMI centile? *Eur J Clin Nutr*. 2005;59(3):419.
- 105. Hayes RJ, Moulton LH. Cluster Randomized Trials 2<sup>nd</sup> Edition. Chapman and Hall/CRC, 2017.
- 106. McNeish D, Stapleton LM. Modeling Clustered Data with Very Few Clusters. *Multivariate Behav Res.* 2016; 51(4): 495-518.
- 107. Gelman A. Bayesian Data Analysis. Chapman and Hall/CRC; 2004; Boca Raton, FL.
- 108. Ma J, Thabane L, Kaczorowski J, Chambers L, Dolvich L, Karwalajtys T, Levitt C. Comparison of Bayesian and Classical Methods in the Analysis of Cluster Randomized Controlled Trials with a Binary Outcome: The Community Hypertension Assessment Trial (CHAT). *BMC Med Res Methodol*. 2009;9:37.
- 109. Spiegelhalter DJ. Bayesian methods for cluster randomized trials with continuous responses. Stat Med. 2001;20 (3): 435-452.
- 110. Gelman A. Prior distributions for variance parameters in hierarchical models. Bayesian Analysis. 2006, 1 (3): 515-533.
- 111. Preacher KJ, Zyphur MJ, Zhang Z. A General Multilevel SEM Framework for Assessing Multilevel Mediation. *Psychol Methods*. 2010;15(3): 209-233.
- 112. Cho SJ, Preacher KJ, Bottge BA. Detecting Intervention Effects in a Cluster-Randomized Design Using Multilevel Structural Equation Modeling for Binary Responses. *Appl Psychol Meas*. 2015;39(8):627-642.
- 113. Muthen LK, Muthen BO. (1998-2017). Mplus User's Guide. Eighth Edition. Los Angeles, CA: Muthen & Muthen.
- 114. Cui Z, Seburg EM, Sherwood NE, Faith MS, Ward DS. Recruitment and retention in obesity prevention and treatment trials targeting minority or low-income children: a review of the clinical trials registration database. *Trials*. 2015 Dec;16(1):564.
- 115. Stekhoven DJ, Buhlmann P. MissForest--non-parametric missing value imputation for mixed-type data. *Bioinformatics*. 2012;28(1):112-118.
- 116. Rubin DB, Schenker N. Multiple imputation in health-care databases: an overview and some applications. *Stat Med.* Apr 1991;10(4):585-598.

117. Casey JA, Savitz DA, Rasmussen SG, Ogburn EL, Pollak J, Mercer DG, Schwartz BS. Unconventional natural gas development and birth outcomes in Pennsylvania, USA. *Epidemiology*. 2016;27(2):163.

- 118. Psek W, Davis FD, Gerrity G, Stametz RA, Bailey-Davis L, Darer J, Henninger D, Sellers D. Leadership perspectives on operationalizing the learning health care system in an integrated delivery system. *EGEMS (Wash DC)*. 2016; 4(3):6.
- 119. Psek WA, Darer J, Stametz R, Bailey-Davis L, Davis D, Faucett WA, Gerrity G, Sellers D, Henninger D. Operationalizing the Learning Health Care System in an Integrated Delivery System. *EGEMS (Wash DC)*. 2015; 3(1):1122.
- 120. Johnson SL, Ryan SM, Kroehl M, Moding KJ, Boles RE, Bellows LL. A longitudinal intervention to improve young children's liking and consumption of new foods: findings from the Colorado LEAP study. *International Journal of Behavioral Nutrition and Physical Activity*. 2019 Dec;16(1):49.
- 121. Kolotourou M, Radley D, Chadwick P, Smith L, Orfanos S, Kapetanakis V, Singhal A, Cole TJ, Sacher PM. Is BMI alone a sufficient outcome to evaluate interventions for child obesity?. *Child Obes*. 2013;9(4):350-6.
- 122. Bailey-Davis L, Virus A, McCoy TA, Wojtanowski A, Vander Veur SS, Foster GD. Middle school student and parent perceptions of government-sponsored free school breakfast and consumption: A qualitative inquiry in an urban setting. *J Acad Nutr Diet*. 2013;113(2):251-7.
- 123. Savage JS, Neshteruk CD, Balantekin KN, Birch LL. Low-Income women's feeding practices and perceptions of dietary guidance: A qualitative study. *Matern Child Health J.* 2016;20(12):2510-7.
- 124. Bailey-Davis L, Hess LB, Marini M, Mowery J, Lutcher S, Savage JS. WIC nutritionist perspectives on opportunities and challenges regarding care coordination with primary care providers for early childhood obesity prevention. *J Patient Cent Res Rev.* 2016 Aug, 3(3):219
- 125. Bailey-Davis L, Poulsen M, Pollak J, Hirsch AG, Glass TA, Schwartz BS. Home food rules in relation to youth eating behaviors, body mass index, waist circumference, and percent body fat. *J Adolesc Health*. 2017 Mar;60(3):270-276. PMID: 27889403.
- 126. Poulsen MN, Knapp E, Pollak J, Hirsch AG, Bailey-Davis L, Schwartz BS. Comparing objective measures of the built environment in their associations with youth physical activity and sedentary behavior across heterogenous geographies. *Health & Place*. 2018 Jan;49:30-38. PMID: 29161656.
- 127. Peyer K, Welk G, Bailey-Davis L, Chen S. County health indicators and obesity rates in Pennsylvania. *BMC Public Health*. 2016 May 14;16(1):404. PMID: 27180170.
- 128. Bailey-Davis L, Peyer KL, Fang Y, Kim JK, Welk GJ. Effects of enhancing school-based body mass index screening reports with parent education on report utility and parental intent to modify obesity risk factors. *Child Obes*. 2017 Apr;13(2):164-171. PMID: 2809904.
- 129. Dzewaltowski DA, Glasgow RE, Klesges LM, Estabrooks PA, Brock E. RE-AIM: evidence-based standards and a Web resource to improve translation of research into practice. *Annals of Behavioral Medicine*. 2004 Oct 1;28(2):75.

- 130. Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. *Health Education Research*. 2006 Aug 31;21(5):688-94.
- 131. Glasgow RE, Klesges LM, Dzewaltowski DA, Bull SS, Estabrooks P. The future of health behavior change research: what is needed to improve translation of research into health promotion practice?. *Annals of Behavioral Medicine*. 2004 Feb 1;27(1):3-12.
- 132. Klesges LM, Dzewaltowski DA, Glasgow RE. Review of external validity reporting in childhood obesity prevention research. *Am J Prev Med*. 2008 Mar 1;34(3):216-23.
- 133. Dzewaltowski DA, Estabrooks PA, Welk G, Hill J, Milliken G, Karteroliotis K, Johnston JA. Healthy youth places: a randomized controlled trial to determine the effectiveness of facilitating adult and youth leaders to promote physical activity and fruit and vegetable consumption in middle schools. *Health Education & Behavior*. 2009 Jun;36(3):583-600.
- 134. Ma X, Barnes TL, Freedman DA, Bell BA, Colabianchi N, Liese AD. Test–retest reliability of a questionnaire measuring perceptions of neighborhood food environment. *Health Place*. 2013;21:65-9.
- 135. Moore LV, Diez Roux AV, Franco M. Measuring availability of healthy foods: agreement between directly measured and self-reported data. *Am J Epidemiol*. 2012;175(10):1037-44.
- 136. Boslaugh SE, Luke DA, Brownson RC, Naleid KS, Kreuter MW. Perceptions of neighborhood environment for physical activity: Is it "who you are" or "where you live?". *J Urban Health*. 2004;81(4):671-81.
- 137. Benzer JK, Young G, Stolzmann K, Osatuke K, Meterko M, Caso A, White B, Mohr DC. The relationship between organizational climate and quality of chronic disease management. *Health Serv Res.* 2011;46(3):691-711.
- 138. Benzer J, Horner M. A meta-analytic integration and test of psychological climate dimensionality. *Human Resource Management*. 2015;54(3):457-82.
- 139. Mohr DC, Benzer JK, Young GJ. Provider workload and quality of care in primary care settings: moderating role of relational climate. *Med care*. 2013:51(1):108-14.
- 140. Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. *Am J Public Health*. 1999;89(8):1231-4.
- 141. Bleich SN, Bandara S, Bennett WL, Cooper LA, Gudzune KA. US health professionals' views on obesity care, training, and self-efficacy. *Am J Prev Med*. 2015;48(4):411-8.
- 142. Bleich SN, Bennett WL, Gudzune KA, Cooper LA. Impact of physician BMI on obesity care and beliefs. *Obesity (Silver Spring)*. 2012;20(5):999-1005.
- 143. Smith MY, Winkel G, Egert J, Diaz-Wionczek M, DuHamel KN. Patient-physician communication in the context of persistent pain: Validation of a modified version of the patients' perceived involvement in care scale. *J Pain Sympton Manage*. 2006;32(1):71-81.

- 144. Schmidt R, Richter R, Brauhardt A, Hiemisch A, Kiess W, Hilbert A. Parental feeding practices in families with children aged 2–13 years: Psychometric properties and child age-specific norms of the German version of the Child Feeding Questionnaire (CFQ). *Appetite*. 2017;109:154-64.
- 145. Koleilat M, Whaley SE. Reliability and validity of food frequency questions to assess beverage and food group intakes among low-income 2-to 4-year-old children. *J Acad Nutr Diet*. 2016;116(6):931-9.
- 146. Bingham D, Collings P, Clemes S, Costa S, Santorelli G, Griffiths P, Barber S. Reliability and validity of the early years physical activity questionnaire (EY-PAQ). *Sports (Basel)*. 2016;4(2):30.
- 147. Carson V, Janssen I. Associations between factors within the home setting and screen time among children aged 0–5 years: a cross-sectional study. *BMC Public Health*. 2012;12(1):539.
- 148. Anderson DR, Field DE, Collins PA, Lorch EP, Nathan JG. Estimates of young children's time with television: a methodological comparison of parent reports with time-lapse video home observation. *Child Dev.* 1985;56 (5):1345-57.
- 149. Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. *Sleep Med.* 2000;1(1):21-32.
- 150. Paul IM, Hohman EE, Loken E, Savage JS, Anzman-Frasca S, Carper P, Marini ME, Birch LL. Mother-infant room-sharing and sleep outcomes in the INSIGHT study. *Pediatrics*. 2017 Jul 1;140(1):e20170122.
- 151. Seligson JL, Huebner ES, Valois RF. Preliminary validation of the brief multidimensional students' life satisfaction scale (BMSLSS). *Social Indicators Research*. 2003 Feb 1;61(2):121-45.
- 152. Schwartz BS, Stewart WF, Godby S, Pollak J, DeWalle J, Larson S, Mercer DG, Glass TA. Body mass index and the built and social environments in children and adolescents using electronic health records. *Am J Prev Med*. 2011;41(4):e17-28.
- 153. Tenenbaum A, Shefer-Averbuch N, Lazar L, Yakobovitch-Gavan M, Phillip M, Oron T. Growth assessment of children during the COVID-19 pandemic-Can we rely on parental measurements? Acta Paediatr. 2021 Nov;110(11):3040-3045. doi: 10.1111/apa.16034. Epub 2021 Jul 27. PMID: 34289178; PMCID: PMC8444654.
- 154. Chai LK, Collins CE, May C, Holder C, Burrows TL. Accuracy of Parent-Reported Child Height and Weight and Calculated Body Mass Index Compared With Objectively Measured Anthropometrics: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Sep 16;21(9):e12532. doi: 10.2196/12532. PMID: 31538954; PMCID: PMC6754693.
- 155. Huybrects et al. Validity of parent-reported weight and height of preschool children measured at home or estiamted without a home measurement: a validation study. BMC Pediatrics 2011: 11:63

156. Gordon NP, Mellor RG. Accuracy of parent-reported information for estimating prevalence of overweight and obesity in a race-ethnically diverse pediatric clinic population aged 3 to 12. BMC Pediatr. 2015 Feb 12;15:5. doi: 10.1186/s12887-015-0320-0. PMID: 25886135; PMCID: PMC4341231.

- 157. Haddad EN, Kojaoghlanian T, Comstock SS. Moving Toward Remote, Parent-Reported Measurements in Pediatric Anthropometrics for Research and Practice. Front Pediatr. 2022 Mar 8;10:838815. doi: 10.3389/fped.2022.838815. PMID: 35350270; PMCID: PMC8957848.
- 158. Wei R, Ogden CL, Parsons VL, Freedman DS, Hales CM. A method for calculating BMI z-scores and percentiles above the 95th percentile of the CDC growth charts. Ann Hum Biol. 2020 Sep;47(6):514-521. doi: 10.1080/03014460.2020.1808065. Epub 2020 Sep 9. PMID: 32901504.
- 159. Freedman DS, Davies AJG, Kompaniyets L, Lange SJ, Goodman AB, Phan TT, Cole FS, Dempsey A, Pajor N, Eneli I, Christakis DA, Forrest CB. A Longitudinal Comparison of Alternatives to Body Mass Index Z-Scores for Children with Very High Body Mass Indexes. J Pediatr. 2021 Aug;235:156-162. doi: 10.1016/j.jpeds.2021.02.072. Epub 2021 Mar 5. PMID: 33676932.
- 160. Ryder JR, Kelly AS, Freedman DS. Metrics Matter: Toward consensus reporting of BMI and weight-related outcomes in pediatric obesity clinical trials. Obesity. 2022; 30(3):571-572.

# **APPENDIX:**

# Appendix A. Family Nutrition and Physical Activity (FNPA Risk Assessment)

| Family Meals | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
|---|---|---|---|---|
| 1. How often does your child eat breakfast, either at home or at school? | 1 | 2 | 3 | 4 |
| 2. How often does your child eat at least one meal a day with at least one other family member? | 1 | 2 | 3 | 4 |
| Family Eating Practices | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
| 3. How often does your child eat while watching TV? [Includes meals or snacks] | 1 | 2 | 3 | 4 |
| 4. How often does your family eat "fast food?" | 1 | 2 | 3 | 4 |
| Food Choices | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
| 5. How often does your family use packaged "readytoeat" foods? [Includes purchased frozen or ontheshelf entrees, often designed to be microwaved] | 1 | 2 | 3 | 4 |
| 6. How often does your child eat fruits and vegetables at meals or snacks? [Not including juice] | 1 | 2 | 3 | 4 |
| Beverage Choices | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
| 7. How often does your child drink soda pop or sweetened beverages? [Includes regular or diet soda pop, KoolAid, SunnyD, Capri Sun, fruit or vegetable juice, caffeinated energy drinks (Monster/Red Bull), Powerade/Gatorade, etc.] | 1 | 2 | 3 | 4 |
| 8. How often does your child drink lowfat milk for meals or snacks? [Includes 1% or skim dairy, flavored, soy, almond, etc.] | 1 | 2 | 3 | 4 |
| Restriction/Reward | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
| 9. How often does your family monitor the amount of candy, chips, and cookies your child eats? | 1 | 2 | 3 | 4 |
| 10. How often does your family use candy, ice cream or other foods as a reward for good behavior? | 1 | 2 | 3 | 4 |
| Screen Time | Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |

| I | I | 1 ! | I |
|---|---|---|---|
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| Never/<br>Almost<br>Never | Sometimes | Often | Very<br>Often/<br>Always |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| | 1 Never/ Almost Never 1 Never/ Almost Never 1 Never/ Almost Never 1 Never/ Almost Never 1 1 Never/ Almost Never 1 1 1 | Never/ Almost Never 1 2 1 2 1 2 Never/ Almost Never 1 2 1 2 | 123Never/Almost NeverSometimes Often123123Never/Almost NeverSometimes Often123Never/Almost NeverSometimes Often123123Never/Almost NeverSometimes Often123Never/Almost NeverSometimes Often123 |

#### Scoring the FNPA

A number of the items on the FNPA are reverse scored with "Very Often/Always" being the less desirable options, so care should be taken when calculating a total score. Additional resources can be found at myfnpa.org and eatright.org. Items to be Reverse Scored (Construct):

- **Family Eating Practices** 3
- 4 **Family Eating Practices**
- 5 **Food Choices**
- 7 **Beverage Choices**
- 10 Restriction/Reward

Encircle Protocol Version 1.21 Version Date: 11/29/2022 IRB #: 2020-0207

#### 13 **Healthy Environment**

#### **Appendix B. Outcomes Table**

We will measure secondary outcomes and potential mediators and moderators of the intervention models' relative effectiveness on obesity including multi-level factors in the community, clinic, and home settings as well as individual-level factors. Factors that will be assessed at the various levels are detailed below brief descriptions and citations indicating psychometric properties of identified measures. Outcomes that are particularly meaningful to patients are identified in green, PCPs in purple, and health care administrators in blue. The total number of items that parents will be asked to respond to vary by data collection time (Telephone survey= 14 items; Baseline= 156 items; 6-month= 79 items; Follow-up= 97 items). PCPs will be asked 56 items at Baseline; 12-month follow-up= 47 items; 24-month maintenance= 47 items. Health Coaches will be asked 53 items at baseline; 12-month follow-up = 44 items; 24-month maintenance = 44 items.

Table 4. Secondary Outcomes, Covariates, Mediating and Moderating Factors on Intervention Effectiveness by Level

| Lei | vel and Factor | Timing | Items | Respondent and Source |
|---|---|---|---|---|
| CO | MMUNITY* | | | |
| 1. | Community Socioeconomic Deprivation <sup>27</sup> (Moderator) Contextual measure derived from a factor analysis of six indicators previously associated with obesity trajectories among children in the Geisinger catchment area | BL | n/a | US Census,<br>American<br>Community<br>Survey |
| 2. | <b>Rurality (Moderator)</b> Density of persons per square mile within counties and communities where clinics are located, and participants reside | BL | n/a | US Census |
| 3. | <b>Parent perception of neighborhood (Moderator)</b> Food access, availability, and quality <sup>135,136</sup> and neighborhood pleasantness and physical activity availability <sup>28,137</sup> | BL | 14 | P-SQ |
| CL | INIC | | | |
| 4. | <b>Organizational Climate</b> <sup>138-140</sup> <b>(Moderator)</b> Shared meaning PCPs attach to PRO measures and the behaviors they see rewarded, supported and expected, specifically related to workflow and relational climate. | BL<br>FU<br>24 mo. | 3 | PCP-SQ, EHR |
| НС | OME | | | |
| 5. | Household Food Security <sup>141</sup> (Secondary Outcome) USDA Food Security Scale short form, which has been validated with diverse populations | BL<br>FU | 6 | P-SQ |
| 6. | WIC, SNAP, HeadStart participation (Covariate) Current enrollment in US food and nutrition education programs | BL | 1 | P-TS |
| 7. | Demographics (Moderator) Household income, access to reliable automobile | BL | 2 | P-TS |
| IN | DIVIDUAL-PRIMARY CARE PROVIDER-HEALTH COACH | | | |
| 8. | <b>Demographics</b> <sup>142,143</sup> <b>(Covariate)</b> Factors that may be associated with provider adoption and effectiveness of intervention components, including specialty, training, experience, biological sex, race/ethnicity, age, self-reported height and weight status | BL | 9 | PCP-SQ |
| 9. | Attitudes, Norms, Perceived Behavioral Control and Intention about Obesity Prevention Intervention <sup>79</sup> (Mediator) Consistent with the Theory of Planned Behavior, PCPs' attitudes, perception of social norms, and perceived behavioral | BL<br>FU<br>24 mo. | 36 | PCP-SQ |

Encircle Protocol Version 1.21 Version Date: 11/29/2022

IRB #: 2020-0207

| | control recording and a hilling to the different state of the state of | | | 1 |
|---|---|---|---|---|
| | control regarding one's ability to modify FNPA risk factors will predict behavioral | | | |
| | intentions and behavioral intentions will predict extent to which PCPs engage in | | | |
| | the intervention | | | 000.00 |
| 10. | Self-efficacy in Preventive Counseling for Obesity <sup>142,143</sup> (Mediator) Training in | BL | 8 | PCP-SQ |
| | and self-efficacy of providing obesity-related prevention and treatment (adapt | FU | | |
| | for pediatrics) | 24 mo. | | |
| | IVIDUAL-PARENT/CAREGIVER | | | |
| 11. | Perceived Involvement in Care <sup>144</sup> (Secondary Outcome) Scale measures parent | BL (pre | 20 | P-SQ |
| | perception of involvement in clinical encounter (adapt for WCV) | or post | | |
| | | WCV), | | |
| | | FU | | |
| 12. | Food Resource Management <sup>23,92</sup> (Secondary Outcome) Validated scales from | BL, | 9 | P-SQ |
| | the Cooking Matters® program assess participants' shopping behaviors and self- | 6 mo., | | |
| | confidence in buying healthy foods and managing food resources | FU | | |
| 13. | <b>Demographics (Covariates)</b> Biological sex, race/ethnicity, age, self-reported | BL | 11 | P-TS |
| | height and weight status, relationship to child, educational level, employment | | | |
| | status | | | |
| 14. | Attitudes, Norms, Perceived Behavioral Control and Intention about Obesity | BL | 25 | P-SQ |
| | Prevention <sup>78</sup> (Mediator) Consistent with the Theory of Planned Behavior, | | | |
| | parents' attitudes, perception of social norms, and perceived behavioral control | | | |
| | regarding FNPA risk factors will predict behavioral intentions and behavioral | | | |
| | intentions will predict extent to which parents engage in the intervention | | | |
| 15. | Parenting Practices <sup>25,145</sup> (Mediator) 5 domains of parenting practices from the | BL | 28 | P-SQ |
| | Child Feeding Questionnaire: parents perceived responsibility for ensuring their | 6 mo., | | |
| | child eats the right types and amounts of food (Responsibility); concern for their | FU | | |
| | child's future or current weight status (Weight Concern); monitoring of their | | | |
| | child's portions, sweet and high fat food intake (Monitoring); pressure they | | | |
| | perceive they must put on their child to make sure he/she eats enough or | | | |
| | finishes all the food on his/her plate (Pressure); and belief that restrictions or | | | |
| | rewards are necessary in their child's diet (Restriction) | | | |
| INC | IVIDUAL-CHILD | | | |
| | Dietary Behaviors <sup>146</sup> (Secondary Outcome) Parent report of the average intake | BL, | 13 | P-SQ |
| . • . | of fruit, vegetable, sugar-sweetened beverages | 6 mo., | | |
| | or many regetable, sugar sweetened berefuges | FU | | |
| 17. | Physical Activity <sup>147</sup> (Secondary Outcome) Parent report of the average daily | BL, | 16 | P-SQ |
| | hours the preschool-age child was moderately to vigorously active | 6 mo., | | |
| | mount the presented age of the was moderately to vigorously detire | FU FU | | |
| 18. | Screen Time148,149 (Secondary Outcome) Parent report of the average daily | BL, | 4 | P-SQ |
| | hours the child spent watching TV, videos, and playing games on TV, computer, | 6 mo., | | |
| | laptop, iPad, smartphones | FU | | |
| 19. | Brief Infant Sleep Questionnare <sup>150</sup> (Secondary Outcome) Parent report of the | BL, | 9 | P-SQ |
| | average amount of daily sleep the child obtained (naps and bedtime) | 6 mo., | 3 | . 50 |
| | are and amount of daily steep the office obtained (haps and beatime) | FU | | |
| 20 | <b>Life Satisfaction</b> <sup>151</sup> (Secondary outcome) Parent report of the child's satisfaction | BL, | 12 | P-SQ |
| _5. | with life using the domain specific and general Student's Life Satisfaction Scale. | FU | 14 | 1-50 |
| 21 | <b>Demographics (Covariates)</b> Biological sex, birthweight, age, race/ethnicity, | BL | n/a | EHR |

<sup>\*</sup>Communities are defined using a mixed definition of place that incorporates minor civil divisions (boroughs, townships) and census tracts within cities. Families will be geocoded to a community based on their residential address.<sup>152</sup>

**Timing**: Baseline (**BL**): Data collected at or near enrollment. Intermediate follow-up period is at 6 months (**6 mo.**). Follow-up (**FU**) period at 12 months following baseline well child visit (allow up to 15 months for scheduling variance); and 24 months for PCPs and Health Coaches to evaluate maintenance

**Items**: Number of questions asked of respondent

**Respondent:** P indicates parent is respondent; **PCP** indicates primary care provider or Health Coach is respondent. **Source:** Secondary data sources are identified. A telephone survey **(TS)** will be used post- consent and prior to baseline well child visit. Electronic health record **(EHR)** will be referenced at baseline well child visit and follow-up. Other variables will be collected by study questionnaire **(SQ)** following the baseline well child visit.

Appendix C. RE-AIM Elements and Planned Assessment, Indicators, and Data Sources

| RE-AIM Elements<br>(Goal) | Measure | Data Source |
|---|---|---|
| Reach (Determine reach and | Evaluate <b>participation rates</b> overall and by subgroups, including the percent of families who consent to each study arm; complete study follow-up; complete PRO measure (Arms 2 and 3); select FNPA topics for discussion with PCP (Arms 2 and 3); and accept referral to Food Care (Arm 3) | Study Records,<br>EHR |
| representativeness of<br>families who participate<br>in intervention arms) | Evaluate <b>representativeness of participating families</b> by comparing characteristics (e.g., child BMI, age, sex, insurance status; parent age and sex; household food security status, rurality) of participants (i.e., those who consent, complete study follow-up, complete PRO measure, select FNPA topics, or attend Food Care) and non-participants | EHR,<br>Parent telephone<br>survey,<br>Study Records |
| Effectiveness<br>(Evaluate intervention<br>arms' impacts on health | Determine <b>effectiveness</b> of intervention arms on primary and secondary outcomes Determine <b>robustness</b> of effectiveness across subgroups (provider type [e.g., | See Outcomes* See Outcomes* |
| behaviors and outcomes) | MD, DO, CRNP, PA-C], household food security status and rurality, parent weight status, child baseline weight status, biological sex and race/ethnicity) Compare attrition by treatment arms and across subgroups | Study Records |
| Adoption – Providers | Determine <b>rate at which providers adopted intervention</b> arms, including the proportion of WCV in which family-centered preventive counseling is documented, by provider; and the proportion of WCV in which PRO measure is utilized, by provider | EHR |
| (Discern whether interventions will translate to new health care settings) | Evaluate <b>representativeness of providers</b> by comparing provider characteristics (e.g., provider type, age, sex, BMI) associated with higher and lower levels of adoption of intervention components (i.e., family-centered preventive counseling, PRO measure utilization) | PCP-Study<br>Questionnaire,<br>Study Records,<br>EHR |
| | Compare characteristics of PCPs who participate in the study versus those who are unwilling/unable to participate | Non-Participant<br>Survey |
| | Determine fidelity to intervention delivery, including percent of eligible participants referred to Food Care (Arm 3); percent of families referred to Food Care that receive Food Care intervention (Arm 3); proportion of participants that attend in-person or virtual grocery store tour and calls (Arm 3) | Study Records,<br>EHR |
| Implementation<br>(Identify implementation<br>barriers; explain reasons<br>for intervention | Report implementation characteristics such as the time needed for PCP training, intervention delivery, the staffing requirements, iPad availability and programming, and information technology programming requirements, anthropometric measurement techniques (assessed by observation) | Study Records |
| effectiveness, or lack thereof) | Identify whether PCP or parent intent to discuss obesity prevention and related attitudes, norms, and self-efficacy explain intervention implementation. | See Outcomes* |
| | Identify implementation strengths and barriers, including PCP self-reported barriers to implementing obesity prevention counseling; parents self-reported barriers to attending Food Care | PCP Study<br>Questionnaire,<br>Food Care Program<br>Records |
| Maintenance | Evaluate adoption over time, including adaptations made to FNPA and Food Care (Cooking Matters, Parent Training Program) to improve sustainability; reevaluate adoption measures 12 months after baseline intervention contact | EHR,<br>Food Care Program<br>Records |
| (Report sustainability of intervention components over time) | Evaluate PRO measure completion rates 12 months after final intervention contact to determine family participation following the study period; proportion of patients that return to the same clinic for their 1-year follow-up WCV | EHR |
| | Evaluate commitment of health system, clinic leadership, and community partner to ongoing implementation of intervention components | Stakeholder<br>discussions |

\*See Appendix B. Outcomes Table